CLINICAL TRIAL: NCT00520195
Title: Stair Instead of Elevator Use at Work: Cardiovascular Primary Preventive Effects on Hospital Employees.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Geneva (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 06-306 (med06-100)
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Last update posted 2007-08-23 (Estimated); Status verified 2007-08

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Physical activity — Climbing stairs instead of taking elevators at worksite during 12 weeks.

SUMMARY:
This is an intervention study which evaluates the cardiovascular primary preventive effects of using stairs instead of elevators at the worksite during a 12-weeks period. We hypothesize that stair-climbing during working hours can meet the daily amount of physical activity recommended by current public health guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* No or little stair-use at work (< 5 stories/day)
* Sedentary lifestyle

Exclusion Criteria:

* Positive answers to the health screening physical activity readiness questionnaire (PAR-Q)
* Part-time employment < 80%
* Absence of more than 2 weeks during the intervention period
* Intention to begin a weight control program
* Medication changes which may influence blood pressure, lipid or glucose metabolism

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2007-03; Study Completion 2007-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Meyer, MD, Principal Investigator — University Hospitals of Geneva
Locations (1):
- University Hospitals of Geneva, Geneva, Switzerland